CLINICAL TRIAL: NCT03440879
Title: The Effect of Androgen Deprivation Therapy on Regulation of Muscle Protein Metabolism and Blood Glucose
Brief Title: Androgen Deprivation Therapy Muscle Protein Metabolism and Blood Glucose
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: University Hospital, Akershus (Other); Oslo University Hospital (Other); Rigshospitalet, Denmark (Other); University of Copenhagen (Other); King's College London (Other)
Responsible Party: Principal Investigator, Truls Raastad, Professor, Norwegian School of Sport Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PROST100
Record Dates: First submitted 2018-02-01; First posted 2018-02-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer; Resistance Exercise; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT group (Experimental): Prostate cancer patients currently receiving androgen deprivation therapy (Zoladex)
  Interventions: Drug: Zoladex
- No-ADT group (No Intervention): Prostate cancer patients without any history of receiving any form of androgen deprivation therapy

INTERVENTIONS:
Drug: Zoladex — Patients currently treated with Zoladex
  Other Names: Androgen deprivation therapy
  Arms: ADT group

SUMMARY:
Prostate cancer (PCa) patients receiving androgen deprivation therapy (ADT) (e.g., Zoladex), experience troublesome side effects during and after treatment (e.g., loss of lean body mass (LBM) and increased fat mass). Although the negative effects of ADT on muscle mass are well documented, the cellular effects of ADT on muscle tissue are still largely unknown, and studies investigating the mechanisms are highly warranted. Furthermore, understanding the cellular mechanisms through which ADT negatively influences muscle mass and glucose metabolism is important so that appropriate measures can be taken to counteract muscle wasting and comorbidities during ADT. Thus, PCa patients on ADT (Zoladex), along with non-ADT treated PCa patients serving as controls, will be invited to participate in this study, that aims to investigate the influence of ADT on the basal muscle protein turnover, as well as the responses to strength training. Secondary aims are to investigate between-group differences in blood glucose and insulin responses following a meal).

DETAILED DESCRIPTION:
Prostate cancer (PCa) patients receiving androgen deprivation therapy (ADT) (e.g., Zoladex), which leads to castrate levels of testosterone, experience troublesome side effects during and after treatment. Commonly reported side effects are loss of lean body mass (LBM) and increased fat mass, as well as impaired glucose- and fat metabolism. Strength training has shown positive effects on LBM in PCa patients on ADT, however, counteracting a substantial LBM loss observed in the control groups seem to account for the intervention effect seen in several of the individual studies. Thus, the real LBM gain following strength training in PCa patients on ADT may be hampered compared to healthy elderly men, but data on this is limited in the literature.

The planned acute recovery study is a continuation of the physical exercise and prostate cancer (PEPC) trial, which was a randomized controlled trial investigating the effects of strength training on body composition, muscle strength, and muscle cellular outcomes during ADT.

Beyond locomotion and activity of daily living, the skeletal muscle tissue plays an important role in glucose metabolism, and impaired glucose uptake to the muscle is associated with diseases such as diabetes mellitus and cardiovascular diseases. In fact, increased levels of fasted blood glucose and insulin have been reported during the first year of ADT. Interestingly, insulin resistance has been noted as early as three months into the treatment. Insulin resistance may, in addition to the increased risk for metabolic comorbidities, also impair the anabolic response in muscles to feeding and exercise. Consequently, the accelerated muscle mass loss, and the potential limited response to strength training might be interlinked to the reduction in insulin sensitivity in PCa patients receiving ADT.

Although the negative effects of ADT on muscle mass are well documented, the cellular effects of ADT on muscle tissue are still largely unknown, and studies investigating the mechanisms are highly warranted. Furthermore, understanding the cellular mechanisms through which ADT negatively influences muscle mass and glucose metabolism is important so that appropriate measures can be taken to counteract muscle wasting and comorbidities during ADT. The present study is designed to address these issues.

PCa patients on ADT (Zoladex), along with non-ADT treated PCa patients serving as controls, will be invited to participate in this study. The aim is to investigate the influence of ADT on the basal muscle protein turnover, as well as the responses to strength training. Furthermore, secondary aims are to investigate between-group differences in blood glucose and insulin responses following a meal).

ELIGIBILITY:
Inclusion criteria

All of the following conditions must apply to the prospective patient at screening prior to participation:

* Histologically verified prostate cancer, and either currently on Zoladex or without any current or no past usage of any ADT
* Between 18 and 75 years of age
* Capable of reading and understanding Norwegian, and able to provide informed consent
* Treating oncologist/ study medical doctor´s (KMR) approval for participation
* Signed informed consent must be obtained and documented according to Good Clinical Practice (GCP), and national/local regulations.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* Routine resistance training (>1 weekly session, last six months)
* Treated with Warfarin, or if seponation of acetylsalicylic acid is not recommended
* Conditions where heavy resistance exercise is contraindicated:

  * Unregulated hypertension
  * Unstable angina pectoris
  * Recent myocardial infarction (<1 year)
  * Cardiac arrhythmia
  * Chronic obstructive pulmonary disease
  * Severe asthma
  * Recent stroke (<1 year)
  * Epilepsy
  * Insulin-dependent diabetes mellitus
  * Unstable bone lesions with increased risk of fractures
* Conditions where patients ability to complete the training sessions is challenged:

  * Uncontrolled pain
  * Severe arthritis
  * Scheduled hip or knee replacement
  * Pathologic fractures last six months
  * Amputations
  * Walker or wheelchair user
* Mentally incompetent conditions:

  * Severe anxiety or depression
  * Dementia
  * Known alcoholism or substance abuse
  * Mentally retarded

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis rate | The muscle biopsy will be collected two hours after the last exercise session.
  The protein synthesis rate will be calculated based on the increased enrichment of deuterium, which will be ingested the week prior to the acute day, in muscle protein isolated from muscle biopsies. Deuterium enrichment is assessed by mass spectrometry.

SECONDARY OUTCOMES:
Muscle cell signalling | Muscle biopsies will be collected on the Acute day. Muscle biopsies obtained 3.5 (baseline biopsy) and 1 hours (post meal) prior to the last exercise session, and 2 hours (post exercise) after the last exercise session will be used
  Changes in the activity of enzymes involved in anabolic- and catabolic signalling, as well as levels of key enzymes related to glucose metabolism, heat shock proteins, and indicators of autophagy capacity, will be analyzed by western blot according to standard operating procedures.
Plasma insulin levels | A fasted blood sample will be collected first thing in the morning at the Acute day. Then again at 15, 30, 45, 60, 75, 90, 105, and 120 minutes post meal and post exercise.
  Will be collected in EDTA vacutainers through venous catheters, centrifuged and serum will be stored at -20ºC for later analysis. When serum from all patients has been collected, insulin levels will be analyzed.
Plasma glucose levels | A fasted blood sample will be collected first thing in the morning at the Acute day. Then again at 15, 30, 45, 60, 75, 90, 105, and 120 minutes post meal and post exercise.
  Will be collected in EDTA vacutainers through venous catheters, centrifuged and serum will be stored at -20ºC for later analysis. When serum from all patients has been collected, glucose levels will be analyzed, along with other hormones and signaling molecules.
Ribosomal RNA | Muscle biopsies will be obtained at the Acute day. Muscle biopsies for ribosomal RNA analysis will be obtained 3.5 hours prior to the last exercise session (baseline) and 2 hours post the last exercise session (post exercise)
  The expression of ribosomal RNAs (including the large subunit; 28S and 5.8S, and the small subunit; 18S) will be assessed by qPCR, to evaluate the translational capacity of the muscle. Also, the acute change in mRNA expression levels of growth factors (e.g. MGF, IGF-1), ubiquitin-proteasome system (e.g. murf-1 and Atrogin-1), genes involved in autophagy (e.g. LC3 and p62), and other testosterone sensitive genes will be analyzed.

OTHER OUTCOMES:
Single muscle fiber myonuclear domain | Muscle biopsies will be obtained at the Acute day. For the single fiber analysis, only baseline biopsies obtained 3.5 hours prior to the last exercise session will be used.
  Single muscle fibers will be isolated from the biopsy specimen. Later, to evaluate if ADT influences the myonuclear domain size, structural analysis, including evaluation for the 3D spatial arrangement of nuclei in relation to myosin content using a unique analysis algorithm applied to confocal images.
Single muscle fiber power analysis | Muscle biopsies will be obtained at the Acute day. For the single fiber analysis, only baseline biopsies obtained 3.5 hours prior to the last exercise session will be used.
  Single muscle fibers will be isolated from the biopsy specimen, membrane-permeabilized and a series of contractile measures will be used to analyse force and velocity (power) following standard protocols.
Single muscle fiber stiffness | Muscle biopsies will be obtained at the Acute day. For the single fiber analysis, only baseline biopsies obtained 3.5 hours prior to the last exercise session will be used.
  Single muscle fibers will be isolated from the biopsy specimen, membrane-permeabilized and stiffness will be analyzed using standard protocols.
The number of capillaries per fiber | Muscle biopsies will be obtained at the Acute day. For the immunohistochemical analysis, only baseline biopsies obtained 3.5 hours prior to the last exercise session will be used.
  The number of capillaries per fiber will be analyzed by immunohistochemistry according to standard procedures, and used as covariates in several analyses
Muscle fiber-type specific cross-sectional area | Muscle biopsies will be obtained at the Acute day. For the immunohistochemical analysis, only baseline biopsies obtained 3.5 hours prior to the last exercise session will be used.
  The baseline fiber-type specific cross-sectional area, the relative fiber type distribution will be analyzed by immunohistochemistry on muscle cryosections according to standard procedures, and used as covariates in several analyses
Myonuclei numbers | Muscle biopsies will be obtained at the Acute day. For the immunohistochemical analysis, only baseline biopsies obtained 3.5 hours prior to the last exercise session will be used.
  The number of myonuclei will be analyzed by immunohistochemistry according to standard procedures, and used as covariates in several analyses
Lean body mass | 1 day
  Total lean body mass will be evaluated by dual x-ray absorptiometry (Lunar iDXA, GE Healthcare, Madison, USA) and will be used as a covariate in several analysis related to glucose metabolism.
Fat mass | 1 day
  Fat mass will be evaluated by dual x-ray absorptiometry (Lunar iDXA, GE Healthcare, Madison, USA), and will be used as a covariate in several analysis related to glucose metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Truls Raastad, Professor, Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No